CLINICAL TRIAL: NCT03713749
Title: Robotic-assisted Esophagectomy vs. Video-Assisted Thoracoscopic Esophagectomy(REVATE) : a Multicenter Open-label Randomized Controlled Trial
Brief Title: Robotic-assisted Esophagectomy vs. Video-Assisted Thoracoscopic Esophagectomy(REVATE) Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Shanghai Chest Hospital (Other); Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201800322A3C601
Record Dates: First submitted 2018-10-11; First posted 2018-10-22 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-03

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Robotic esophagectomy; Video-assisted thoracoscopic esophagectomy; Recurrent laryngeal nerve lymh node; Esophageal squamous cell carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot Esophagectomy (RE) (Experimental): Patients in the RE group will receive robotic-assisted esophagectomy with standard total two-field lymphadenectomy.
  Interventions: Device: Robot esophagectomy (RE)
- Video-assisted thoracoscopic esophagectomy (VATE) (No Intervention): Patients in the VATE group will receive thoracoscopic esophagectomy with standard total two-field lymphadenectomy.

INTERVENTIONS:
Device: Robot esophagectomy (RE) — Patients in RE group will receive Robotic-assisted surgery in thoracic phase.
  Arms: Robot Esophagectomy (RE)

SUMMARY:
The investigators will assess the adequacy of nodal dissection along the recurrent laryngeal nerve performed with robot-assisted versus video-assisted thoracoscopic esophagectomy in patients with esophageal squamous cell carcinoma through a prospective multicentre randomized study design.

DETAILED DESCRIPTION:
Radical lymph node dissection (LND) along the recurrent laryngeal nerve (RLN) is surgically demanding and can be associated with substantial postoperative morbidity. The question as to whether robot-assisted esophagectomy (RE) might be superior to video-assisted thoracoscopic esophagectomy (VATE) for performing LND along the RLN in patients with esophageal squamous cell carcinoma (ESCC) remains open.

The investigators will conduct a multicenter, open-label, randomized controlled trial (termed REVATE) enrolling patients with ESCC scheduled to undergo LND along the RLN. Patients will be randomly assigned to either RE or VATE. The primary outcome measure will be the rate of unsuccessful LND along the left RLN, which will be defined as 1) failure to remove lymph nodes along the left RLN or 2) occurrence of left RLN palsy following LND. Secondary outcomes will include the number of successfully removed RLN nodes, postoperative recovery, length of hospital stay, 30- and 90-day mortality, quality of life, and oncological outcomes.

ELIGIBILITY:
Inclusion criteria

1. Age between 18~80
2. Histologically proven primary intrathoracic esophageal squamous cell carcinoma and will undergo McKeown MIE and bilateral RLN LND.
3. Patients should have a performance status 0, 1 or 2 according to the European Clinical Oncology Group.
4. Surgical resectable(cT1~4a, N0~3, M0)
5. Written informed consent

Exclusion criteria are

1. Previous major thoracic surgery rendering minimal invasive approach unfeasible
2. prognosis determining malignancy other than esophageal cancer, inability to undergo curative resection and/or follow-up
3. inability to provide oral or written informed consent.
4. pre-existed vocal cord dysfunction will also be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2018-10-22 (Actual); Primary Completion 2022-04-22 (Estimated); Study Completion 2022-12-22 (Estimated)

PRIMARY OUTCOMES:
Rate of unsuccessful LND along the left RLN | Till 6 months postoperatively
  Regardless of the presence of hoarseness, vocal cord function will be assessed by an experienced otolaryngologist using a nexile laryngoscope within one week of surgery. RLN palsy will be classified according to the following variables: site (unilateral versus bilateral); duration (temporary [i.e., recovering within 6 months] versus permanent [i.e. not recovering within 6 months]); and type of treatment required (type I: no therapy required; type II: injury requiring an elective surgical procedure; type III: injury requiring an urgent surgical procedure)

SECONDARY OUTCOMES:
The number of nodes removed along the right and left RLN | The pathological analysis will be finished within 2 weeks.
  number of lymph node removed
Post esophagectomy pneumonia rate | Duration of hospital stay, an expected average of 2~3 weeks
  Post esophagectomy pneumonia is defined according to the Revised Uniform Pneumonia Score which includes temperature[°C](Range ≥ 36.1 and ≤ 38.4 =0, ≤ 36.0 and ≥ 38.5=1); leukocyte count [×1000/uL](≥ 4.0 and ≤ 11.0=0, <4.0 or >11.0=1); and pulmonary radiography(Range No infiltrate=0, Diffused or patchy infiltrate=1, Well-circumscribed infiltrate=2). A sum score of 2 points or higher, of which at least 1 point is assigned because of infiltrative findings on pulmonary radiography, indicates the presence of pneumonia.
Rate of major postoperative complication | Duration of hospital stay, an expected average of 2~3 weeks
  Complication grade: modified Clavien-Dindo classification (MCDC) grade 2-4 Major complications (MCDC grade 2-4) Including: myocardial infarction, anastomotic leakage (clinical or radiologic diagnosis), anastomotic stenosis, chylothorax (chylous leakage, presence of chylous in chest tubes or indication start medium chain triglycerides containing tube feeding, gastric tube necrosis (proven by gastroscopy), pulmonary embolus, deep vein thrombosis.
  Minor complications (MCDC grade 1) Including: wound infections, pleural effusions, delayed gastric emptying
In hospital, 30 day and 90 day mortality | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks and within 30 days or 90 days
  Death occurred during the same hospitalization , within 30 and 90 days after surgery
R0 resection rate | The pathological analysis will be finished within 2 weeks.
  Microscopically negative proximal/distal and circumferential margin
Operation time(thoracic phase) | Day of surgery
  thoracic phase operation time(minutes)
Operation time(abdominal) | Day of surgery
  abdominal phase operation time(minutes)
Total operation time | Day of surgery
  total surgical time (expressed in minutes)
Unexpected events and complications occurring during surgery | Day of surgery, up to 24 hours after surgery.
  massive hemorrhage, perforation of other organs
Blood loss during surgery | Day of surgery, up to 24 hours after surgery.
  blood loss during surgery (expressed in mL per phase)
Rate of thoracotomy conversion | Day of surgery, up to 24 hours after surgery.
  Number of patients requiring conversion to thoracotomy and related reasons
Length of mechanical ventilator use after surgery | Participants will be followed for the duration of hospital stay, an expected average of 2~3 weeks
  expressed in minutes
Length of intensive care unit stay after surgery | Participants will be followed for the duration of hospital stay, an expected average of 2~3 weeks
  expressed in hours
Length of postoperative hospital stay | Participants will be followed for the duration of hospital stay, an expected average of 2~3 weeks
  expressed in days , calculated from the date of surgery to date of discharge
Re-intubation rate | Participants will be followed for the duration of hospital stay, an expected average of 2~3 weeks
  Need for re-intubation after extubation
Re-entry ICU rate | Participants will be followed for the duration of hospital stay, an expected average of 2~3 weeks
  Need to transfer back from ward to ICU after surgery
Overall survival rate | Assessed 24/36/60 months after surgery
  From date of surgery until the date of death from any cause
Disease free survival rate | Assessed up to 24/36/60 months after surgery
  From date of surgery until the date of first documented recurrence
Hospital Anxiety and Depression Scale (HADS) | pre-operative < 5 days and 4 weeks, 3/6 months and yearly up to 5 years post-operatively.
  The HADS aims to measure symptoms of anxiety and depression and consists of 14 items,seven items for the anxiety subscale and seven for the depression subscale. The questionnaire responses were analysed in the light of the results of this estimation of the severity of both anxiety and of depression. This enabled a reduction of the number of items in the questionnaire to just seven reflecting anxiety and seven reflecting depression.(Of the seven depression items five reflected aspects of reduction in pleasure response). Each item had been answered by the patient on a four point (0-3) response category so the possible scores ranged from 0 to 21 for anxiety and 0 to 21 for depression. a score of 0 to 7 for either subscale could be regarded as being in the normal range, a score of 11 or higher indicating probable presence ('caseness') of the mood disorder and a score of 8 to 10 being just suggestive of the presence of the respective state.
European Organisation for Research and Treatment of Cancer(EORTC) QLQ-C30 , QLQ-OES18 | pre-operative < 5 days and 4 weeks, 3/6 months and yearly up to 5 years post-operatively.
  The EORTC QLQ-C30 incorporates a range of QOL issues in five functional scales (physical, role, cognitive, emotional, and social), three symptom scales (fatigue, pain, and nausea/vomiting), a global health/QOL scale, and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The EORTC QLQ-OES18 contains four symptom scales (dysphagia, eating disorders, reflux, and pain) and six single items (difficulty swallowing saliva, choking, dry mouth, taste disorder, cough, and speech-related issues). Each question has four response choices ranging from 1 (not at all) to 4 (very much), except for the global QOL scale, which has seven response options ranging from 1 (very poor) to 7 (excellent). All questionnaire responses are linearly transformed to scores from 0 to 100.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung memorial hospital-Linkou, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Udagawa H, Ueno M, Shinohara H, Haruta S, Kaida S, Nakagawa M, Tsurumaru M. The importance of grouping of lymph node stations and rationale of three-field lymphoadenectomy for thoracic esophageal cancer. J Surg Oncol. 2012 Nov;106(6):742-7. doi: 10.1002/jso.23122. Epub 2012 Apr 13. PMID 22504922
- [Background] Mizutani M, Murakami G, Nawata S, Hitrai I, Kimura W. Anatomy of right recurrent nerve node: why does early metastasis of esophageal cancer occur in it? Surg Radiol Anat. 2006 Aug;28(4):333-8. doi: 10.1007/s00276-006-0115-y. Epub 2006 May 23. PMID 16718401
- [Background] Sato Y, Kosugi S, Aizawa N, Ishikawa T, Kano Y, Ichikawa H, Hanyu T, Hirashima K, Bamba T, Wakai T. Risk Factors and Clinical Outcomes of Recurrent Laryngeal Nerve Paralysis After Esophagectomy for Thoracic Esophageal Carcinoma. World J Surg. 2016 Jan;40(1):129-36. doi: 10.1007/s00268-015-3261-8. PMID 26464155
- [Background] Fujita H, Sueyoshi S, Tanaka T, Fujii T, Toh U, Mine T, Sasahara H, Sudo T, Matono S, Yamana H, Shirouzu K. Optimal lymphadenectomy for squamous cell carcinoma in the thoracic esophagus: comparing the short- and long-term outcome among the four types of lymphadenectomy. World J Surg. 2003 May;27(5):571-9. doi: 10.1007/s00268-003-6913-z. Epub 2003 Apr 28. PMID 12715226
- [Background] Gockel I, Kneist W, Keilmann A, Junginger T. Recurrent laryngeal nerve paralysis (RLNP) following esophagectomy for carcinoma. Eur J Surg Oncol. 2005 Apr;31(3):277-81. doi: 10.1016/j.ejso.2004.10.007. PMID 15780563
- [Background] Berry MF, Atkins BZ, Tong BC, Harpole DH, D'Amico TA, Onaitis MW. A comprehensive evaluation for aspiration after esophagectomy reduces the incidence of postoperative pneumonia. J Thorac Cardiovasc Surg. 2010 Dec;140(6):1266-71. doi: 10.1016/j.jtcvs.2010.08.038. Epub 2010 Sep 29. PMID 20884018
- [Background] Hulscher JB, van Sandick JW, Devriese PP, van Lanschot JJ, Obertop H. Vocal cord paralysis after subtotal oesophagectomy. Br J Surg. 1999 Dec;86(12):1583-7. doi: 10.1046/j.1365-2168.1999.01333.x. PMID 10594510
- [Background] Luketich JD, Pennathur A, Awais O, Levy RM, Keeley S, Shende M, Christie NA, Weksler B, Landreneau RJ, Abbas G, Schuchert MJ, Nason KS. Outcomes after minimally invasive esophagectomy: review of over 1000 patients. Ann Surg. 2012 Jul;256(1):95-103. doi: 10.1097/SLA.0b013e3182590603. PMID 22668811
- [Background] Zhou C, Zhang L, Wang H, Ma X, Shi B, Chen W, He J, Wang K, Liu P, Ren Y. Superiority of Minimally Invasive Oesophagectomy in Reducing In-Hospital Mortality of Patients with Resectable Oesophageal Cancer: A Meta-Analysis. PLoS One. 2015 Jul 21;10(7):e0132889. doi: 10.1371/journal.pone.0132889. eCollection 2015. PMID 26196135
- [Background] Biere SS, van Berge Henegouwen MI, Maas KW, Bonavina L, Rosman C, Garcia JR, Gisbertz SS, Klinkenbijl JH, Hollmann MW, de Lange ES, Bonjer HJ, van der Peet DL, Cuesta MA. Minimally invasive versus open oesophagectomy for patients with oesophageal cancer: a multicentre, open-label, randomised controlled trial. Lancet. 2012 May 19;379(9829):1887-92. doi: 10.1016/S0140-6736(12)60516-9. Epub 2012 May 1. PMID 22552194
- [Background] Noshiro H, Iwasaki H, Kobayashi K, Uchiyama A, Miyasaka Y, Masatsugu T, Koike K, Miyazaki K. Lymphadenectomy along the left recurrent laryngeal nerve by a minimally invasive esophagectomy in the prone position for thoracic esophageal cancer. Surg Endosc. 2010 Dec;24(12):2965-73. doi: 10.1007/s00464-010-1072-4. Epub 2010 May 22. PMID 20495981
- [Background] Park SY, Kim DJ, Yu WS, Jung HS. Robot-assisted thoracoscopic esophagectomy with extensive mediastinal lymphadenectomy: experience with 114 consecutive patients with intrathoracic esophageal cancer. Dis Esophagus. 2016 May;29(4):326-32. doi: 10.1111/dote.12335. Epub 2015 Feb 26. PMID 25716873
- [Background] van der Sluis PC, Ruurda JP, Verhage RJ, van der Horst S, Haverkamp L, Siersema PD, Borel Rinkes IH, Ten Kate FJ, van Hillegersberg R. Oncologic Long-Term Results of Robot-Assisted Minimally Invasive Thoraco-Laparoscopic Esophagectomy with Two-Field Lymphadenectomy for Esophageal Cancer. Ann Surg Oncol. 2015 Dec;22 Suppl 3:S1350-6. doi: 10.1245/s10434-015-4544-x. Epub 2015 May 29. PMID 26023036
- [Background] Cerfolio RJ, Wei B, Hawn MT, Minnich DJ. Robotic Esophagectomy for Cancer: Early Results and Lessons Learned. Semin Thorac Cardiovasc Surg. 2016 Spring;28(1):160-9. doi: 10.1053/j.semtcvs.2015.10.006. Epub 2015 Oct 30. PMID 27568155
- [Background] Suda K, Ishida Y, Kawamura Y, Inaba K, Kanaya S, Teramukai S, Satoh S, Uyama I. Robot-assisted thoracoscopic lymphadenectomy along the left recurrent laryngeal nerve for esophageal squamous cell carcinoma in the prone position: technical report and short-term outcomes. World J Surg. 2012 Jul;36(7):1608-16. doi: 10.1007/s00268-012-1538-8. PMID 22392356
- [Background] Weksler B, Sharma P, Moudgill N, Chojnacki KA, Rosato EL. Robot-assisted minimally invasive esophagectomy is equivalent to thoracoscopic minimally invasive esophagectomy. Dis Esophagus. 2012 Jul;25(5):403-9. doi: 10.1111/j.1442-2050.2011.01246.x. Epub 2011 Sep 7. PMID 21899652
- [Background] Chao YK, Hsieh MJ, Liu YH, Liu HP. Lymph Node Evaluation in Robot-Assisted Versus Video-Assisted Thoracoscopic Esophagectomy for Esophageal Squamous Cell Carcinoma: A Propensity-Matched Analysis. World J Surg. 2018 Feb;42(2):590-598. doi: 10.1007/s00268-017-4179-0. PMID 28801820
- [Background] Low DE, Alderson D, Cecconello I, Chang AC, Darling GE, D'Journo XB, Griffin SM, Holscher AH, Hofstetter WL, Jobe BA, Kitagawa Y, Kucharczuk JC, Law SY, Lerut TE, Maynard N, Pera M, Peters JH, Pramesh CS, Reynolds JV, Smithers BM, van Lanschot JJ. International Consensus on Standardization of Data Collection for Complications Associated With Esophagectomy: Esophagectomy Complications Consensus Group (ECCG). Ann Surg. 2015 Aug;262(2):286-94. doi: 10.1097/SLA.0000000000001098. PMID 25607756
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Background] van der Sluis PC, Ruurda JP, van der Horst S, Verhage RJ, Besselink MG, Prins MJ, Haverkamp L, Schippers C, Rinkes IH, Joore HC, Ten Kate FJ, Koffijberg H, Kroese CC, van Leeuwen MS, Lolkema MP, Reerink O, Schipper ME, Steenhagen E, Vleggaar FP, Voest EE, Siersema PD, van Hillegersberg R. Robot-assisted minimally invasive thoraco-laparoscopic esophagectomy versus open transthoracic esophagectomy for resectable esophageal cancer, a randomized controlled trial (ROBOT trial). Trials. 2012 Nov 30;13:230. doi: 10.1186/1745-6215-13-230. PMID 23199187
- [Background] Li ZG, Zhang XB, Wen YW, Liu YH, Chao YK. Incidence and Predictors of Unsuspected Recurrent Laryngeal Nerve Lymph Node Metastases After Neoadjuvant Chemoradiotherapy in Patients with Esophageal Squamous Cell Carcinoma. World J Surg. 2018 Aug;42(8):2485-2492. doi: 10.1007/s00268-018-4516-y. PMID 29380005
- [Background] Chiu CH, Wen YW, Chao YK. Lymph node dissection along the recurrent laryngeal nerves in patients with oesophageal cancer who had undergone chemoradiotherapy: is it safe? Eur J Cardiothorac Surg. 2018 Oct 1;54(4):657-663. doi: 10.1093/ejcts/ezy127. PMID 29608683
- [Background] Rice TW, Ishwaran H, Ferguson MK, Blackstone EH, Goldstraw P. Cancer of the Esophagus and Esophagogastric Junction: An Eighth Edition Staging Primer. J Thorac Oncol. 2017 Jan;12(1):36-42. doi: 10.1016/j.jtho.2016.10.016. Epub 2016 Oct 31. PMID 27810391
- [Background] Japan Esophageal Society. Japanese Classification of Esophageal Cancer, 11th Edition: part I. Esophagus. 2017;14(1):1-36. doi: 10.1007/s10388-016-0551-7. Epub 2016 Nov 10. No abstract available. PMID 28111535
- [Background] Weijs TJ, Seesing MF, van Rossum PS, Koeter M, van der Sluis PC, Luyer MD, Ruurda JP, Nieuwenhuijzen GA, van Hillegersberg R. Internal and External Validation of a multivariable Model to Define Hospital-Acquired Pneumonia After Esophagectomy. J Gastrointest Surg. 2016 Apr;20(4):680-7. doi: 10.1007/s11605-016-3083-5. Epub 2016 Feb 16. PMID 26883435
- [Background] Tachimori Y, Ozawa S, Numasaki H, Matsubara H, Shinoda M, Toh Y, Udagawa H, Fujishiro M, Oyama T, Uno T; Registration Committee for Esophageal Cancer of the Japan Esophageal Society. Efficacy of lymph node dissection by node zones according to tumor location for esophageal squamous cell carcinoma. Esophagus. 2016;13:1-7. doi: 10.1007/s10388-015-0515-3. Epub 2015 Nov 17. PMID 26752982
- [Derived] Chao YK, Li Z, Jiang H, Wen YW, Chiu CH, Li B, Shang X, Fang TJ, Yang Y, Yue J, Zhang X, Zhang C, Liu YH. Multicentre randomized clinical trial on robot-assisted versus video-assisted thoracoscopic oesophagectomy (REVATE trial). Br J Surg. 2024 Jul 2;111(7):znae143. doi: 10.1093/bjs/znae143. PMID 38960881
- [Derived] Chao YK, Li ZG, Wen YW, Kim DJ, Park SY, Chang YL, van der Sluis PC, Ruurda JP, van Hillegersberg R. Robotic-assisted Esophagectomy vs Video-Assisted Thoracoscopic Esophagectomy (REVATE): study protocol for a randomized controlled trial. Trials. 2019 Jun 10;20(1):346. doi: 10.1186/s13063-019-3441-1. PMID 31182150